CLINICAL TRIAL: NCT01201382
Title: Depression Prevention Initiative - A Study of IPT-AST in School Settings
Brief Title: Depression Prevention Initiative - A Study of Interpersonal Psychotherapy-Adolescent Skills Training (IPT-AST) in School Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Rutgers University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MH087481; R01MH087481 (NIH)
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Depression
Keywords: Depression; Prevention; Adolescents
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IPT-AST (Experimental): Interpersonal Psychotherapy-Adolescent Skills Training
  Interventions: Behavioral: IPT-AST
- Group Counseling (Active Comparator): Group Counseling
  Interventions: Behavioral: Group Counseling

INTERVENTIONS:
Behavioral: IPT-AST — A school-based group prevention program that includes 2 individual pre-group sessions, 8 weekly 90 minute group sessions, an individual mid-group session and 4 booster sessions
  Other Names: Interpersonal Psychotherapy-Adolescent Skills Training
  Arms: IPT-AST
Behavioral: Group Counseling — Usual group counseling as delivered by school counselors; 1 pre-group session, 1 mid-group session, 8 90-minute group sessions, 4 booster sessions
  Other Names: Usual group counseling
  Arms: Group Counseling

SUMMARY:
This study is a randomized controlled trial comparing Interpersonal Psychotherapy-Adolescent Skills Training (IPT-AST) to group counseling (GC) for the prevention of depression in adolescents. The project will: (1) identify adolescents with elevated depressive symptoms but who do not meet criteria for a current mood disorder diagnosis; (2) randomize eligible adolescents to either IPT-AST (N = 100) or GC (N = 100); (3) assess depressive symptoms, depressive disorders, global functioning, interpersonal functioning, comorbid conditions and school related indices at baseline, mid-intervention, post-intervention, and at 6-, 12-, 18-, and 24-month follow-up; (4) examine the effects of IPT-AST on depression and various domains of functioning at each time point; and (5) conduct analyses to examine potential mediators and moderators of the association between IPT-AST and depression outcomes. This study will yield data on the efficacy of IPT-AST relative to GC for the prevention of depressive symptoms and depressive disorders. It will also provide information about the mechanisms of action of IPT-AST and determine for whom IPT-AST is most effective.

ELIGIBILITY:
Inclusion Criteria:

* In 7th-10th grades at intake
* Center for Epidemiologic Studies Depression Scale(CES-D) Score > 16
* At least 2 symptoms on the K-SADS depression section (score of 2 or 3), one of which is either depressed mood, irritability, or anhedonia
* Adolescent must be English-speaking
* Parent speaks English or Spanish

Exclusion Criteria:

* CES-D Score < 15
* Fewer than 2 depression symptoms on the K-SADS (score of 2 or 3) or 2 or more symptoms on the K-SADS with no report of depressed mood, irritability, or anhedonia
* Suicide attempt or self-mutilation in the past year, current active suicidal ideation, and/or history of a clinically significant suicidal behavior (i.e., with intent to die and high medical lethality) or repeated patterns of self-injurious behavior
* Presence of current Major Depressive Disorder, dysthymia, substance abuse, schizophrenia, bipolar disorder, conduct disorder, or psychosis

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 185 (Actual)
Dates: Start 2010-10; Primary Completion 2015-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Presence of a Major Depressive Episode, Dysthymia or Depressive Disorder Not Otherwise Specified (NOS) on the Schedule for Affective Disorders for School Aged Children - Present and Life Time Version (K-SADS-PL) | Post intervention (approximately 3 months post baseline)
  Presence of a depression diagnosis as measured by a semi-structured diagnostic evaluation
Presence of a Major Depressive Episode, Dysthymia or Depressive Disorder NOS on the K-SADS-PL | 6-months post-intervention
Presence of a Major Depressive Episode, Dysthymia or Depressive Disorder NOS on the K-SADS-PL | 12-months post-intervention
Presence of a Major Depressive Episode, Dysthymia or Depressive Disorder NOS on the K-SADS-PL | 18-months post-intervention
Presence of a Major Depressive Episode, Dysthymia or Depressive Disorder NOS on the K-SADS-PL | 24-months post-intervention

SECONDARY OUTCOMES:
Children's Depression Rating Scale-Revised (CDRS-R) | Post intervention (approximately 3 months after baseline)
  Scores on the CDRS-R
Children's Depression Rating Scale-Revised | 6-months post-intervention
Children's Depression Rating Scale-Revised | 12-months post-intervention
Children's Depression Rating Scale-Revised | 18-months post-intervention
Children's Depression Rating Scale-Revised | 24 months post-intervention
Children's Global Assessment Scale (CGAS) | Post intervention (approximately 3 months following baseline)
  Assesses global functioning
Children's Global Assessment Scale | 6-months post-intervention
Children's Global Assessment Scale | 12-months post-intervention
Children's Global Assessment Scale | 18-months post-intervention
Children's Global Assessment Scale | 24-months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jami F Young, Ph.D., Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Rutgers University, Piscataway, New Jersey
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

DOCUMENTS (1):
  • Informed Consent Form (2011-04-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT01201382/ICF_000.pdf